CLINICAL TRIAL: NCT03340168
Title: Kinetic Time Courses of Bisphenol-S in Female Volunteers Orally and Dermally Exposed to Bisphenol-S
Brief Title: Kinetic Time Courses of Bisphenol-S in Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Michèle Bouchard, Full professor, Université de Montréal
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EST-17-174
Record Dates: First submitted 2017-11-07; First posted 2017-11-13 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: PHARMACOKINETICS
Keywords: Bisphenol S, toxicokinetics
MeSH Terms: interventions — bisphenol S

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bisphenol-S kinetics - oral exposure (Experimental): Six female volunteers will be exposed orally acute at the reference dose level(0.1 mg / kg bw). For the administration, the product will be dissolved in ethanol (100 mg / ml equivalent to 10 mg / 100 μl) and the solution will be deposited on a cookie (deposit of about 70 μl of solution on a cookie for an individual of 70 kg) and the ethanol is allowed to evaporate before giving each volunteer, with the subsequent consumption of 100 ml of water.
  Interventions: Other: Bisphenol-S
- Bisphenol-S kinetics - dermal exposure (Experimental): volunteers will be exposed dermally acute at a dose of 1 mg / kg bw. The solution will be applied to an area of 40 cm2 of the forearm and delimited by the indelible marker. The BPS will be added in suspension in an aqueous solution containing 1% of carboxymethylcellulose and administered in the form of drops (70 .mu.l for an individual of 70 kg). The treated area will be left uncoated and unwashed for a period of 4 hours. After 4 hours, the application area will be washed with water and soap. This type of application is therefore similar to an exposure of the general population via the skin (manipulation of cash receipts).
  Interventions: Other: Bisphenol-S

INTERVENTIONS:
Other: Bisphenol-S — Oral and dermal exposure in volunteers

SUMMARY:
The time course of bisphenol S in plasma and urine will be monitored in female adults exposed to a single oral and dermal dose of bisphenol-S. Six female will be recruited. Blood and urine will be collected at specified times post-treatment. Bisphenol concentrations will be measured in those samples.

DETAILED DESCRIPTION:
As a first step, volunteers will be exposed orally acutely to 0.1 mg / kg of body weight (bw) orally (corresponding to 7 mg for an individual of 70 kg). According to the recent assessment by the US Environmental Protection Agency (U.S. EPA), this dose is considered to be associated with no adverse effect for a subchronic exposure scenario in rats (EPA, 2014). The deuterated form of bisphenol S (BPS d8, Toronto Research Chemical) will be used to avoid potential interference with BPS in the diet. The dose that will be administered to volunteers (0.1 mg / kg bw) orally, in deuterated form, is identical to that previously used in a study in volunteers exposed to Bisphenol A (0.1 mg / kg of BPA-d6 administered oral in volunteers) (Thayer et al., 2015).

The BPS reference dose (RfD) was established based on a 45-day parental toxicity study in orally exposed male rats with No-Observed Adverse Effect Level (NOAEL) 10 mg / kg bw (Lowest-Observed-Adverse-Effect-Level (LOAEL) of 60 mg / kg bw / day for parental toxicity, and a NOAEL and LOAEL value of 60 and 300 mg / kg bw / day for reproductive toxicity) (EPA 2014) (page 4-282). The dose administered in volunteers will be 100 times lower than the NOAEL and consider an inter-species uncertainty factor of 10 and interindividual of 10. The six volunteers will then be exposed orally acutely to the previously determined dose (0.1 mg / kg bw).

For the administration, the product will be dissolved in ethanol (100 mg / ml equivalent to 10 mg / 100 μl) and the solution will be deposited on a cookie (deposit of about 70 μl of solution on a cookie for an individual of 70 kg) and the ethanol is allowed to evaporate before giving each volunteer, with the subsequent consumption of 100 ml of water.

In a second component, volunteers will be exposed dermally acute at a dose of 1 mg / kg bw. It is important to note that there is currently no recommended reference dose for dermal exposure. Studies on the toxicokinetics of bisphenol A (BPA) in the animal and human model estimated that the absorption fraction was 8.6 ± 2.1% in human skin explants (n = 7) (Demierre et al. , 2012). The expected dermal administration dose assumes that dermal absorption is <10% based on the Demierre study and therefore may be higher than the oral dose. Preliminary experience on a volunteer will be done before doing all the planned volunteers.

About 48 hours before dermal exposure to BPS, it is recommended to remove the hair on the forearm while taking care not to irritate the skin too much. The solution will then be applied to an area of 40 cm2 of the forearm and delimited by the indelible marker. The BPS will be added in suspension in an aqueous solution containing 1% of carboxymethylcellulose and administered in the form of drops (70 µl for an individual of 70 kg). The treated area will be left uncoated and unwashed for a period of 4 hours. After 4 hours, the application area will be washed with water and soap. This type of application is therefore similar to an exposure of the general population via the skin (manipulation of cash receipts).

The kinetics of bisphenol S (BPS) and its metabolite (glucurono-conjugated BPS (BPSG) in blood will be documented by collecting blood by venous puncture at time: -30 min (control sample) and at fixed times during a 48-h period post-treatment: at 15 min, 30 min, 45 min, 1 h, 1 h 15, 1 h 30, 1 h 45, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 24 h and 48 h post-treatment (n = 17 samples per individual). A catheter will be inserted during the day of exposure, to allow serial blood sampling. A total of 20 ml will be collected per time point, which represent a total of 340 ml, which is inferior to a blood donation.

To document urinary time cours, complete urine voids will be collectedin distinct bottles at fixed time periods: -10 h-0 h (control) and 0-2 h, 2-4 h, 4-6 h, 6-8 h, 8-10 h, 10-12 h, 12-14 h, 14-24 h, 24-48 h and 48-72 h post-administration (n = 11 collections per individual and all void between two time points will be pooled).

ELIGIBILITY:
Inclusion Criteria:

* Female

Exclusion Criteria:

* People with liver or kidney problems or cancer

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Toxicokinetics of bisphenol-S | 0-72 h post-treatment
  Time course in blood and urine

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Bouchard, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No